CLINICAL TRIAL: NCT04386720
Title: Measurement of Airway Opening Pressure (AOP) in Patients With Acute Respiratory Distress Syndrom With Pressure Volume Curve on the Ventilator and With Electrical Impedance Tomography (EIT) Derived Method in Comparison of the Curves in Patients With or Without Covid 19 Pneumoniae.
Brief Title: Measurement of Airway Opening Pressure (AOP) in Patients With Acute Respiratory Distress Syndrom and With or Without Covid 19.
Acronym: POVA-TIE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/15
Record Dates: First submitted 2020-05-11; First posted 2020-05-13 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Ventilation Induced Lung Injury; Airway Closer; Airway Opening Pressure; Electrical Impedance Tomography; Pressure Volume curve
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mechanical ventilation in ARDS requires protective ventilation and PEEP. Airway closer has to be overcome to reduce lung heterogeneity, AOP is measured globally with a ventilator PV curve without PEEP. EIT derived PV curve is another method that could determine heterogeneity of AOP between both lung.

This study aims to determine whether AOP measured with EIT derived PV curve is similar to AOP on the ventilator PV curve and see if AOP is different between lungs.

If airway closer is higher on one lung, global AOP on the ventilator PV curve probably estimates the other lung.

DETAILED DESCRIPTION:
Scientific justification:

In one third of Acute Respiratory Distress Syndrome (ARDS), tidal inflation starts when an airway opening pressure (AOP) is overcome 1. This phenomenon of airway closure has been underestimated and misinterpreted. Recent research demonstrates that airway closure is a matter of concern as it participates to the heterogeneity of tidal ventilation distribution and it can amplify Ventilator Induced Lung Injury (VILI). The detection of airway closure and the measurement of AOP need a pressure volume curve at low flow and no positive end expiratory pressure (PEEP). However, this will measure a global AOP whereas ventilation is heterogeneous between the two lungs in ARDS. EIT is an interesting monitoring tool that could allow EIT derived PV curve construction with measurement of regional AOP2, right vs left lung. The investigor wants to compare global AOP on ventilator PV curve with left and right lung EIT derived AOP measurements. Recent Covid 19 pneumoniae is responsible for numerous acute respiratory distress with severe hypoxemia. Phenotypes are discussed with differences in terms of respiratory mechanics. It is therefore important to describe specifically Covid 19 patients with ARDS.

Strategy description:

Patients with moderate to severe ARDS equipped with EIT will be included. PEEP will be titrated with PEEP-EIT method. A classical low flow PV curve from without PEEP will be done, the acquisition of EIT data during PV curve will be analysed secondary with a dedicated software. PV curve on the ventilator will be analysed to determine if there is an airway closer phenomenon. Reconstruction of EIT derived PV curve will determine, first: if there is a left and/or right lung airway closer phenomenon, and second: the value of each lung AOP.

Follow up description:

* Measurement of ventilator pressures, flow and volume before/during/after the PV curve.
* Last chest X Ray and arterial blood gases,
* Haemodynamic data.

ELIGIBILITY:
* Inclusion criteria:

  - Patients hospitalized in the ICU and who suffered moderate to severe ARDS (Berlin criteria) equipped EIT over the age of 18.
* Exclusion criteria:

  * Broncho-pleural leaks
  * ECMO
  * Pregnant or breastfeeding woman.
  * Guardianship or curatorship
  * Deprived of liberty
  * No health insurance
  * Impossibility to correctly position the EIT belt (e.g., dressings, chest drainage, etc.)
  * Contra indications to EIT (e.g., implantable cardiac defibrillator, pacemaker, instable spinal lesions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients hospitalized in thoracic intensive care of Haut-Lévêque Hospital, with moderate to severe ARDS according to the Berlin criteria.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Comparison of the PV curves | At inclusion day
  global ventilator method vs regional EIT derived method in all patients

SECONDARY OUTCOMES:
Comparison of regional AOP | At inclusion day
  Global ventilator method vs regional EIT derived method in regional AOP, right and left lungs
Comparison of the different AOPs with the level of PEEP | At inclusion day
  Comparison selected by the EIT-PEEP method

CONTACTS AND LOCATIONS:
Locations (1):
- HOPITAL HAUT-LEVEQUE - Service Réanimation thoracique, Pessac, France